CLINICAL TRIAL: NCT01440881
Title: Does Nesiritide Provide Renal Protection By Attenuating the Inflammatory Response
Brief Title: Does Nesiritide Provide Renal Protection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 70-2010; 09KW-03 (Other Grant/Funding Number: Florida Department of Health)
Record Dates: First submitted 2011-02-10; First posted 2011-09-27 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Renal Failure
Keywords: renal failure; cardiopulmonary bypass
MeSH Terms: conditions — Renal Insufficiency | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nesiritide (Active Comparator): infuses at 0.01 MCG (micrograms)/KG (kilograms)/min (minute) for 48 hours
  Interventions: Drug: Nesiritide
- Placebo (Placebo Comparator): infuses at 0.01MCG/KG/min for 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nesiritide — infuses at 0.01MCG/KG/min for 48 hours
  Other Names: kidney protection post cardiopulmonary bypass.
  Arms: Nesiritide
Drug: Placebo — infuses at 0.01MCG/KG/min for 48 hours
  Other Names: kidney protection post cardiopulmonary bypass
  Arms: Placebo

SUMMARY:
This project evaluates whether nesiritide, human recombinant brain natriuretic peptide, confers renal protection during cardiovascular surgery by attenuating the inflammatory response.

DETAILED DESCRIPTION:
This will be a randomized, prospective blinded pilot study comparing nesiritide to placebo in patients undergoing aortic arch, ascending aorta, aortic valve or mitral valve surgery with baseline GFR 30-90ml/min. Patients were randomized to either placebo or nesiritide (administered prophylactically starting in the operating room prior to incision at 0.01 mcg/kg /minute with no bolus and continued for 48 hours).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery on their aortic arch, ascending aorta, or having aortic valve or mitral valve surgery
* Baseline MDRD (modification of diet in renal disease) calculated GFR (Glomerular Filtration Rate) 30-90 ml/min.
* Signed Informed Consent

Exclusion Criteria:

* Age <18 or >80
* Ejection Fraction <30%.
* Presence of endocarditis or other infection.
* Presence or anticipated use of an intra-aortic balloon pump.
* History of an organ transplant.
* History of an adverse reaction to nesiritide.
* Surgery performed without cardiopulmonary bypass.
* Receiving Aprotinin
* Dopamine administered in doses <5 mcg /kg min.
* Women of child bearing potential or pregnant or breastfeeding.
* Participation in any other investigational trial
* Jehovah Witness
* Bleeding Disorder
* Active Endocarditis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Beaver, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Starting in June 2010 and ending in December 2012, subjects were seen in outpatient clinics or in the hospital. The pre-operative labs were used to screen and enroll subjects.
Pre-assignment Details: Out of the 37 signed informed consent there were 8 subjects who were consented and did not participate: 2 subjects changed their mind, 5 subjects creatinine level was not within the protocol level for participation, 1 subject surgery was canceled. This left 29 subjects to participate in the study.
Groups:
- Nesiritide: infuses at 0.01 micrograms (MCG)/kilograms (KG)/minute (min) for 48 hours
  Nesiritide: infuses at 0.01MCG/KG/min for 48 hours
- Placebo: infuses at 0.01micrograms (MCG)/kilograms (KG)/minute (min) for 48 hours
  Placebo: infuses at 0.01MCG/KG/min for 48 hours
Period: Overall Study
Arm/Group | Nesiritide | Placebo
Started | 14 | 15
Completed | 14 | 14
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nesiritide | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 13
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Measure Neutrophils to Measure Kidney Injury
Description: 0.35 mL of whole blood from each patient was applied to a microfluidics chip to isolate neutrophils. Total RNA was subsequently isolated and gene expression (for all genes listed below) was measured with an Affymetrix gene chip. Data was normalized using RMA (Robust multi-array average) and expressed as log2 expression.
Time Frame: 30 days from the start of infusion
Measure: Mean (Standard Deviation); unit: log2 expression
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 14 | 15
log2 expression
  Gene: TUFT1 | 5.453 (0.251) | 5.630 (0.195)
  Gene: IL23A | 4.508 (0.177) | 4.546 (0.301)
  Gene: C6orf145 | 5.501 (0.216) | 5.444 (0.156)
  Gene: HIST1H1C | 8.888 (0.506) | 9.404 (0.903)
  Gene: TBC1D26 /// ZNF286A | 4.990 (0.092) | 4.930 (0.113)
  Gene: RPL27 | 9.269 (0.191) | 9.315 (0.214)
  Gene: LOC440087 | 3.553 (0.181) | 3.647 (0.218)
  Gene: PRAMEF8 | 5.828 (0.232) | 5.856 (0.233)
  Gene: RPL26 | 7.440 (0.205) | 7.481 (0.212)
  Gene: OXT | 6.899 (0.175) | 6.884 (0.102)
  Gene: GIPC3 | 6.158 (0.124) | 6.097 (0.114)
  Gene: ZNF540 | 4.284 (0.110) | 4.255 (0.120)
  Gene: FAM98C | 6.778 (0.146) | 6.857 (0.129)
  Gene: PTOV1 | 8.234 (0.210) | 8.153 (0.149)
  Gene: RPS16 | 9.077 (0.195) | 9.012 (0.221)
  Gene: ERCC1 | 5.798 (0.171) | 5.843 (0.242)
  Gene: LOC339344 | 7.522 (0.238) | 7.502 (0.164)
  Gene: ATG10 | 5.347 (0.390) | 5.286 (0.308)
  Gene: SLC35C1 | 6.422 (0.155) | 6.358 (0.188)
  Gene: PTPMT1 /// NDUFS3 /// PTPMT1 | 6.702 (0.168) | 6.706 (0.177)
  Gene: SIDT2 | 6.792 (0.215) | 6.870 (0.161)
  Gene: Q6ZVY8_HUMAN | 5.229 (0.124) | 5.132 (0.214)
  Gene: CECR5 | 5.519 (0.108) | 5.499 (0.105)
  Gene: VPS35 | 9.042 (0.339) | 8.974 (0.379)
  Gene: LGALS2 | 5.513 (0.174) | 5.565 (0.187)
  Gene: NDUFA6 | 6.496 (0.334) | 6.680 (0.455)
  Gene: LOC497190 /// NP_001011880.1 | 6.469 (0.089) | 6.470 (0.116)
  Gene: CXorf52 | 6.151 (0.480) | 6.301 (0.387)
  Gene: MAP4K4 | 10.656 (0.121) | 10.651 (0.159)
  Gene: LOC441241 /// VKORC1L1 | 6.418 (0.349) | 6.533 (0.453)
  Gene: DBF4 | 4.706 (0.245) | 4.776 (0.364)
  Gene: SP100 | 9.074 (0.242) | 9.205 (0.191)
  Gene: TPT1 | 9.177 (0.139) | 9.242 (0.125)
  Gene: LOC285908 | 7.517 (0.173) | 7.454 (0.322)
  Gene: LOXHD1 | 6.886 (0.336) | 6.742 (0.398)
  Gene: DYM | 8.158 (0.241) | 8.088 (0.281)
  Gene: Q6ZU44_HUMAN | 4.953 (0.200) | 4.751 (0.159)
  Gene: BAZ2B | 8.802 (0.330) | 8.811 (0.117)
  Gene: GRM8 | 4.303 (0.114) | 4.259 (0.142)
  Gene: Q6ZP42_HUMAN | 4.967 (0.251) | 5.040 (0.336)
  Gene: HTR2B | 4.337 (0.263) | 4.037 (0.289)
  Gene: PRSS3 | 6.338 (0.123) | 6.241 (0.118)
  Gene: LOC728449 /// ANXA8L2 | 5.755 (0.105) | 5.801 (0.195)
  Gene: RPS24 | 7.029 (0.153) | 7.063 (0.153)
  Gene: DOLPP1 | 5.707 (0.218) | 5.759 (0.200)
  Gene: UBQLN1 | 9.129 (0.174) | 9.172 (0.214)
  Gene: TNFSF15 | 5.080 (0.296) | 5.072 (0.330)
  Gene: Q5QFB9_HUMAN | 4.770 (0.456) | 4.430 (0.427)
  Gene: CYP19A1 | 3.696 (0.126) | 3.725 (0.131)
  Gene: Q6UWF5_HUMAN | 3.851 (0.309) | 3.893 (0.209)
  Gene: LOC340204 /// NP_001010886.1 | 4.453 (0.208) | 4.437 (0.273)
  Gene: CCDC76 | 3.702 (0.211) | 3.627 (0.211)

2. Primary Outcome: The Examine and Measure Cytokines to Measure Kidney Injury
Description: Serial measurement of serum cytokine profiles were measured with multiplex Luminex plates that enable the simultaneous measurement of 23 cytokines.
Time Frame: 30 days from the start of infusion
Population: randomized per protocol
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Placebo: infuses at 0.01 MCG (micrograms)/KG (kilograms)/min (minute) for 48 hours Placebo: infuses at 0.01MCG/KG/min for 48 hours
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 14 | 15
pg/ml
  IL-6 baseline | 1.750 [0.407 to 7.189] | 1.959 [0.433 to 9.273]
  IL-6 time point 0 | 28.167 [18.008 to 40.283] | 63.930 [49.471 to 99.201]
  IL-6 1 hour post bypass | 33.457 [24.237 to 48.103] | 57.412 [40.169 to 120.589]
  IL-6 2 hour post bypass | 44.383 [35.629 to 62.855] | 43.523 [35.380 to 118.481]
  IL-6 4hour post bypass | 35.759 [30.562 to 72.392] | 37.967 [27.729 to 78.084]
  IL-6 6 hour post bypass | 28.593 [24.190 to 52.719] | 27.840 [19.707 to 56.711]
  IL-6 8 hours post bypass | 29.794 [21.559 to 46.560] | 21.673 [14.773 to 44.934]
  IL-6 24 hours post bypas | 29.513 [20.704 to 35.399] | 34.650 [24.828 to 41.952]
  IL8 baseline | 5.377 [3.554 to 10.042] | 5.238 [2.621 to 9.596]
  IL-8 0 time point | 16.821 [13.256 to 31.274] | 18.962 [13.751 to 35.247]
  IL8- 1 hour post bypass | 17.107 [14.959 to 23.696] | 20.873 [14.384 to 42.450]
  IL8-2 hour post bypass | 17.068 [15.574 to 34.241] | 23.607 [14.957 to 36.670]
  IL8 4 hour post bypass | 16.005 [14.241 to 23.305] | 17.627 [15.373 to 26.853]
  IL8 6 hour post bypass | 14.290 [12.090 to 23.910] | 19.880 [12.237 to 24.394]
  IL8 8hour post bypass | 14.550 [11.221 to 19.530] | 16.282 [9.661 to 19.578]
  IL8 24 hour post bypass | 12.264 [9.647 to 16.549] | 14.600 [10.591 to 16.596]
  IL10 baseline | 8.063 [2.930 to 23.735] | 9.130 [8.056 to 14.720]
  IL10 0 time point | 1289.776 [665.231 to 1691.249] | 2206.177 [1666.118 to 2748.541]
  IL 10 1 hour post bypass | 1558.903 [1169.255 to 2519.783] | 2074.906 [1196.237 to 2482.497]
  IL10 2 hour post bypass | 667.765 [549.079 to 918.143] | 844.352 [406.264 to 1097.627]
  IL 10 4 hour post bypass | 309.351 [213.114 to 450.841] | 230.101 [134.756 to 470.378]
  IL 10 6 hour post bypass | 107.778 [81.076 to 231.203] | 95.925 [81.336 to 262.041]
  IL 10 8 hour post bypass | 103.791 [70.919 to 174.660] | 84.070 [65.525 to 93.980]
  IL 10 24 hour post bypass | 18.597 [10.610 to 29.888] | 34.862 [23.830 to 44.290]
  TNF alpha baseline | 6.286 [4.961 to 7.346] | 5.402 [3.009 to 8.012]
  TNF alpha 0 time point | 8.253 [6.526 to 9.649] | 7.795 [5.688 to 11.360]
  TNF alpha 1hour post bypass | 10.729 [9.265 to 12.630] | 13.310 [8.519 to 15.580]
  TNF alpha 2 hour post bypass | 9.855 [8.885 to 11.307] | 11.729 [9.975 to 13.947]
  TNF alpha 4 hour post bypass | 8.843 [7.002 to 13.359] | 9.291 [6.509 to 13.568]
  TNF alpha 6 hour post bypass | 7.185 [5.607 to 11.008] | 7.953 [4.840 to 10.815]
  TNF alpha 8 hour post bypass | 5.175 [4.284 to 8.931] | 5.212 [2.800 to 6.250]
  TNF alpha 24 hour post bypass | 4.620 [1.971 to 6.091] | 4.525 [3.365 to 6.618]
  TNF beta baseline | 1.162 [0.000 to 7.714] | 0.056 [0.000 to 1.623]
  TNF beta 0 time point | 1.110 [0.055 to 8.519] | 0.000 [0.000 to 1.031]
  TNF beta 1 hour post bypass | 0.898 [0.000 to 8.648] | 0.000 [0.000 to 0.338]
  TNF beta 2 hour post bypass | 1.302 [0.198 to 6.717] | 0.406 [0.000 to 0.950]
  TNF beta 4 hour post bypass | 1.698 [0.518 to 5.051] | 0.074 [0.000 to 0.706]
  TNF beta 6 hour post bypass | 1.234 [0.149 to 5.796] | 0.219 [0.000 to 0.498]
  TNF beta 8 hour post bypass | 1.389 [0.198 to 4.883] | 0.058 [0.000 to 1.199]
  TNF beta 24 hour post bypass | 0.309 [0.000 to 8.662] | 0.404 [0.000 to 1.589]
  VEGF baseline | 102.054 [41.148 to 151.786] | 44.971 [33.233 to 78.745]
  VEGF 0 time point | 70.647 [27.779 to 121.082] | 35.773 [28.314 to 57.292]
  VEGF 1 hour post bypass | 89.814 [48.225 to 157.629] | 48.928 [20.450 to 67.083]
  VEGF 2 hour post bypass | 91.881 [50.242 to 153.212] | 41.695 [22.994 to 93.293]
  VEGF 4 hour poswt bypass | 88.005 [43.210 to 161.897] | 30.529 [19.981 to 68.473]
  VEGF 6 hour post bypass | 83.581 [42.650 to 144.648] | 26.226 [24.178 to 56.900]
  VEGF 8 hour post bypass | 84.494 [39.215 to 137.660] | 36.577 [28.953 to 70.361]
  VEGF 24 hour post bypass | 76.771 [43.973 to 121.778] | 64.660 [29.898 to 98.724]
  MCP-1 baseline | 174.848 [143.677 to 215.191] | 182.708 [146.434 to 250.832]
  MCP-1 0 timepoint | 478.742 [381.513 to 650.308] | 455.129 [315.690 to 678.396]
  MCP-1 1 hour post bypass | 483.095 [408.870 to 822.554] | 572.955 [429.401 to 955.947]
  MCP-1 2 hour post bypass | 441.203 [318.854 to 709.902] | 502.992 [429.098 to 912.456]
  MCP-1 4 hour post bypass | 265.736 [211.247 to 432.764] | 325.249 [288.906 to 392.275]
  MCP-1 6 hour post bypass | 191.735 [168.518 to 310.851] | 218.561 [195.837 to 311.979]
  MCP-1 8 hour post bypass | 180.749 [128.801 to 232.952] | 177.527 [149.096 to 239.253]
  MCP-1 24 hour post bypass | 202.621 [159.322 to 236.815] | 215.708 [162.058 to 247.327]
  EGF baseline | 47.564 [28.196 to 75.165] | 39.794 [26.826 to 74.659]
  EGF 0 timepoint | 31.242 [14.718 to 69.982] | 21.983 [15.145 to 47.203]
  EGF 1 hour post bypass | 35.745 [21.122 to 79.986] | 19.395 [14.549 to 33.210]
  EGF 2 hour post bypass | 24.052 [17.339 to 56.405] | 23.662 [12.757 to 29.182]
  EGF 4 hour post bypass | 29.841 [15.028 to 48.199] | 19.141 [11.353 to 23.873]
  EGF 6 hour post bypass | 33.050 [15.711 to 44.114] | 22.655 [15.988 to 28.370]
  EGF 8 post bypass | 27.022 [12.558 to 47.269] | 26.093 [16.129 to 36.236]
  EGF 24 hour post bypass | 30.494 [13.189 to 63.895] | 17.768 [15.228 to 54.487]
  IL-1 alpha baseline | 12.372 [4.209 to 26.931] | 2.754 [0.938 to 17.260]
  IL-1 alpha 0 time | 41.216 [20.491 to 49.241] | 31.597 [15.750 to 32.969]
  IL-1 alpha 1 hour post bypass | 26.101 [10.389 to 43.738] | 21.069 [8.055 to 29.453]
  IL-1 alpha 2 hour post bypass | 22.122 [12.403 to 36.620] | 17.803 [6.430 to 25.311]
  IL-1 alpha 4 hour post bypass | 18.137 [14.394 to 25.199] | 10.732 [3.549 to 17.785]
  IL-1 alpha 6 hour post bypass | 15.148 [7.747 to 24.294] | 5.745 [2.233 to 16.900]
  IL-1 alpha 8 hour post bypass | 9.334 [4.901 to 21.816] | 5.376 [1.093 to 10.690]
  IL-1 alpha 24 hour post bypass | 2.974 [1.426 to 19.918] | 1.389 [0.000 to 9.465]
  IL-1Beta baseline | 1.014 [0.000 to 2.938] | 0.394 [0.000 to 1.227]
  IL-1Beta 0 time point | 0.775 [0.000 to 2.599] | 0.492 [0.000 to 0.775]
  IL-1Beta 1 hour post bypass | 0.653 [0.015 to 3.005] | 0.430 [0.000 to 1.252]
  IL-1Beta 2 hour post bypass | 1.311 [0.001 to 3.051] | 0.450 [0.000 to 1.411]
  IL-1Beta 4 hour post bypass | 1.716 [0.155 to 2.256] | 0.310 [0.000 to 1.349]
  IL-1Beta 6 hour post bypass | 1.119 [0.000 to 2.531] | 0.366 [0.000 to 1.237]
  IL-1Beta 8 hour post bypass | 0.875 [0.000 to 2.022] | 0.462 [0.000 to 0.946]
  IL-1Beta 24 hour post bypass | 0.000 [0.000 to 1.876] | 0.170 [0.000 to 1.742]
  IL-1RA baseline | 26.419 [0.000 to 33.138] | 0.000 [0.000 to 21.347]
  IL-1RA 0 time point | 41.945 [14.544 to 96.153] | 53.721 [24.312 to 108.171]
  IL-1RA 1 hour post bypass | 68.792 [13.478 to 112.704] | 71.444 [35.659 to 163.338]
  IL-1RA 2 hour post bypass | 98.089 [65.649 to 227.339] | 237.080 [104.788 to 396.803]
  IL-1RA 4 hour post bypass | 105.861 [48.931 to 173.007] | 152.630 [90.576 to 330.576]
  IL-1RA 6 hour post bypass | 67.705 [31.982 to 141.879] | 75.226 [30.186 to 128.904]
  IL-1RA 8 hour post bypass | 45.097 [3.338 to 70.559] | 27.442 [14.928 to 120.969]
  IL-1RA 24 hour post bypass | 21.181 [0.00 to 38.018] | 15.765 [0.000 to 38.997]
  IL-2 baseline | 0.850 [0.027 to 3.993] | 0.068 [0.000 to 1.008]
  IL-2 0 timepoint | 1.130 [0.126 to 3.741] | 0.401 [0.000 to 1.189]
  IL-2 1 hour post bypass | 1.714 [0.069 to 3.466] | 0.059 [0.000 to 1.352]
  IL-2 2 hour post bypass | 1.714 [0.430 to 4.723] | 1.110 [0.054 to 2.040]
  IL-2 4 hour post bypass | 1.753 [0.685 to 3.601] | 0.870 [0.086 to 1.939]
  IL-2 6 hour post bypass | 1.297 [0.215 to 3.952] | 0.923 [0.045 to 1.433]
  IL-2 8 hour post bypass | 1.281 [0.198 to 2.792] | 0.599 [0.030 to 1.271]
  IL-2 24 hour post bypass | 0.921 [0.000 to 2.495] | 0.172 [0.000 to 1.039]
  IL-3 baseline | 0.093 [0.000 to 0.552] | 0.000 [0.000 to 0.292]
  IL-3 0 timepoint | 0.185 [0.000 to 0.544] | 0.000 [0.000 to 0.196]
  IL-3 1 hour post bypass | 0.000 [0.000 to 0.410] | 0.000 [0.000 to 0.200]
  IL-3 2 hour post bypass | 0.000 [0.000 to 0.355] | 0.000 [0.000 to 0.258]
  IL-3 4 hour post bypass | 0.000 [0.000 to 0.372] | 0.000 [0.000 to 0.191]
  IL_3 6 hour post bypass | 0.061 [0.000 to 0.377] | 0.000 [0.000 to 0.217]
  IL-3 8 hour post bypass | 0.061 [0.000 to 0.293] | 0.000 [0.000 to 0.199]
  IL_3 24 hour post bypass | 0.073 [0.000 to 0.445] | 0.000 [0.000 to 0.234]
  IL-4 baseline | 4.295 [0.717 to 19.395] | 0.166 [0.000 to 2.459]
  IL-4 0 timepoint | 6.285 [0.084 to 10.721] | 0.359 [0.000 to 1.944]
  IL-4 1 hour post bypass | 6.221 [1.321 to 12.502] | 0.414 [0.000 to 2.437]
  IL_4 2 hour post bypass | 5.534 [3.030 to 10.564] | 1.381 [0.139 to 3.258]
  IL-4 4 hour post bypass | 6.743 [1.647 to 10.309] | 0.958 [0.000 to 3.584]
  IL-4 6 hour post bypass | 4.859 [2.256 to 8.644] | 0.746 [0.000 to 2.877]
  IL-4 8 hour post bypass | 4.063 [1.329 to 7.170] | 0.000 [0.000 to 2.378]
  IL_4 24 hour post bypass | 3.634 [0.000 to 8.419] | 0.000 [0.000 to 1.864]
  IL-5 baseline | 0.563 [0.000 to 4.234] | 0.353 [0.000 to 1.233]
  IL-5 0 timepoint | 0.134 [0.000 to 0.808] | 0.016 [0.000 to 0.580]
  IL-5 1 hour post bypass | 0.169 [0.000 to 1.145] | 0.040 [0.000 to 0.789]
  IL-5 2 hour post bypass | 0.291 [0.000 to 0.901] | 0.000 [0.000 to 1.104]
  IL-5 4 hour post bypass | 0.626 [0.000 to 1.089] | 0.016 [0.000 to 1.083]
  IL-5 6 hour post bypass | 0.334 [0.000 to 1.252] | 0.210 [0.000 to 0.900]
  IL-5 8 hour post bypass | 0.387 [0.020 to 0.574] | 0.431 [0.000 to 0.796]
  IL-5 24 hour post bypass | 0.373 [0.000 to 1.366] | 0.503 [0.055 to 0.794]
  IL-7 baseline | 4.032 [3.525 to 4.584] | 2.987 [1.617 to 3.672]
  IL-7 0 timepoint | 3.673 [2.620 to 6.634] | 4.311 [2.539 to 5.931]
  IL-7 1 hour post bypass | 2.973 [2.000 to 4.488] | 1.822 [1.483 to 4.524]
  IL-7 2 hour post bypass | 2.469 [1.965 to 4.588] | 2.104 [1.187 to 4.430]
  IL-7 4 hour post bypass | 3.061 [2.245 to 4.719] | 2.530 [1.377 to 3.134]
  IL-7 6 hour post bypass | 3.391 [2.527 to 4.717] | 2.317 [1.509 to 3.027]
  IL-7 8 hour post bypass | 3.506 [1.769 to 4.277] | 2.354 [1.655 to 4.597]
  IL-7 24 hour post bypass | 3.656 [0.000 to 4.629] | 4.097 [1.163 to 5.022]
  IL-13 baseline | 0.922 [0.000 to 11.185] | 0.000 [0.000 to 2.027]
  IL-13 0 timepoint | 0.133 [0.000 to 4.913] | 0.000 [0.000 to 0.302]
  IL-13 1 hour post bypass | 0.719 [0.000 to 5.817] | 0.000 [0.000 to 0.989]
  IL-13 2 hour post bypass | 2.352 [0.000 to 4.561] | 1.185 [0.000 to 1.794]
  IL-13 4 hour post bypass | 1.571 [0.000 to 3.443] | 0.287 [0.000 to 1.029]
  IL-13 6 hour post bypass | 1.138 [0.000 to 5.160] | 0.000 [0.000 to 0.746]
  IL-13 8 hour post bypass | 0.786 [0.000 to 2.603] | 0.000 [0.000 to 0.573]
  IL-13 24 hour post bypass | 0.094 [0.000 to 5.222] | 0.000 [0.000 to 1.233]
  IL-15 baseline | 1.905 [0.810 to 6.231] | 0.969 [0.000 to 2.795]
  IL-15 0 timepoint | 3.200 [1.493 to 6.739] | 3.093 [1.483 to 3.914]
  IL-15 1 hour post bypass | 4.228 [2.920 to 7.884] | 3.981 [3.016 to 6.153]
  IL-15 2 hour post bypass | 5.556 [2.814 to 8.172] | 4.641 [3.381 to 6.860]
  IL-15 4 hour post bypass | 5.723 [4.258 to 7.128] | 4.423 [3.542 to 6.768]
  IL-15 6 hour post bypass | 5.021 [3.049 to 7.138] | 4.395 [3.004 to 5.526]
  IL-15 8 hour post bypass | 4.984 [2.873 to 6.096] | 3.316 [1.841 to 3.989]
  IL-15 24 hour post bypass | 6.120 [4.023 to 6.695] | 4.996 [3.434 to 6.161]
  IL-17 baseline | 1.171 [0.000 to 2.730] | 0.000 [0.000 to 2.552]
  IL-17 0 time point | 0.765 [0.000 to 4.558] | 0.117 [0.000 to 0.943]
  IL-17 1 hour post bypass | 2.174 [0.202 to 7.780] | 0.130 [0.000 to 0.768]
  IL-17 2 hour post bypass | 1.381 [0.475 to 7.394] | 0.456 [0.000 to 1.228]
  IL-17 4 hour post bypass | 1.682 [0.412 to 3.982] | 0.000 [0.000 to 1.899]
  IL-17 6 hour post bypass | 0.815 [0.196 to 3.582] | 0.162 [0.000 to 1.290]
  IL- 17 8 hour post bypass | 0.817 [0.000 to 2.857] | 0.000 [0.000 to 1.574]
  IL-17 24 hour post bypass | 0.397 [0.000 to 3.457] | 0.0000 [0.000 to 2.480]
  IP-10 baseline | 506.657 [490.553 to 713.745] | 475.656 [304.609 to 527.253]
  IP-10 0 time point | 2340.935 [1691.645 to 3585.567] | 1790.035 [1554.647 to 3807.319]
  IP-10 1 hour post bypass | 1828.152 [1293.335 to 2297.526] | 2298.747 [1478.354 to 2763.464]
  IP-10 2 hour post bypass | 1571.877 [1105.554 to 1991.710] | 1365.169 [961.057 to 1998.178]
  IP-10 4 hour post bypass | 1072.023 [910.335 to 1338.142] | 855.843 [608.726 to 1465.772]
  IP-10 6 hour post bypass | 704.208 [579.992 to 775.662] | 575.429 [396.859 to 1059.186]
  IP-10 8 hour post bypass | 448.938 [292.341 to 570.529] | 449.376 [295.222 to 675.398]
  IP-10 24 hour post bypass | 243.332 [213.669 to 265.925] | 241.467 [157.583 to 333.628]
  MIP-1 alpha baseline | 2.251 [0.000 to 4.082] | 0.000 [0.000 to 3.064]
  MIP-1 alpha 0 time point | 8.880 [5.954 to 11.191] | 10.109 [4.705 to 14.815]
  MIP-1 alpha 1 hour post bypass | 9.042 [7.056 to 17.518] | 9.182 [6.161 to 18.698]
  MIP-1 alpha 2 hour post bypass | 6.610 [5.410 to 8.129] | 6.268 [4.309 to 10.444]
  MIP-1 alpha 4 hour post bypass | 4.024 [1.888 to 7.931] | 4.309 [0.462 to 4.872]
  MIP-1 alpha 6 hour post bypass | 3.017 [0.154 to 6.573] | 0.870 [0.000 to 2.779]
  MIP-1 alpha 8 hour post bypass | 1.933 [0.000 to 5.446] | 0.000 [0.000 to 3.036]
  MIP-1 alpha 24 hour post bypass | 1.279 [0.000 to 2.870] | 0.000 [0.000 to 1.806]
  MIP-1 beta baseline | 22.626 [19.968 to 33.454] | 18.167 [14.254 to 23.434]
  MIP-1 beta 0 time point | 55.229 [41.784 to 105.270] | 47.617 [35.620 to 55.731]
  MIP-1 beta 1 hour post bypass | 85.082 [60.080 to 159.731] | 57.405 [48.300 to 71.806]
  MIP-1 beta 2 hour post bypass | 53.750 [38.134 to 86.942] | 40.900 [34.678 to 48.173]
  MIP-1 beta 4 hour post bypass | 34.010 [24.951 to 44.472] | 24.018 [22.720 to 28.116]
  MIP-1 beta 6 hour post bypass | 26.524 [21.681 to 52.531] | 20.263 [17.094 to 25.972]
  MIP-1 beta 8 hour post bypass | 22.676 [17.226 to 37.256] | 18.522 [16.173 to 24.292]
  MIP-1 beta 24 hour post bypass | 18.726 [15.327 to 23.802] | 16.082 [12.354 to 20.734]
  G-CSF baseline | 50.953 [31.490 to 81.650] | 43.984 [24.558 to 51.463]
  G-CSF 0 time point | 92.559 [66.615 to 120.739] | 150.567 [117.980 to 180.159]
  G-CSF 1 hour post bypass | 124.298 [76.047 to 150.769] | 253.527 [176.006 to 281.092]
  G-CSF 2 hour post bypass | 249.816 [176.392 to 280.874] | 297.668 [206.217 to 439.136]
  G-CSF 4 hour post bypass | 285.277 [210.293 to 373.804] | 311.452 [215.692 to 576.031]
  G-CSF 6 hour post bypass | 252.546 [193.625 to 305.081] | 224.425 [197.557 to 382.366]
  G-CSF 8 hour post bypass | 264.061 [161.506 to 298.064] | 243.292 [175.307 to 312.665]
  G-CSF 24 hour post bypass | 309.690 [161.764 to 385.424] | 199.849 [128.946 to 286.537]

3. Primary Outcome: The Examine and Measure Endothelin-1 to Measure Kidney Injury
Description: Serial measurements of Endothelin-1 levels were measured to determine if natriuretic peptides exert their renal protective effects by preserving renal afferent arteriole flow by antagonizing the vasoconstrictive effects of Endothelin-1.
Time Frame: 30 days from the start of infusion
Population: randomized as outlined in the protocol
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 14 | 15
pg/ml
  baseline prior to infusion | 1.778 [1.443 to 2.149] | 1.239 [0.991 to 2.557]
  time point 0 | 2.096 [1.899 to 2.568] | 2.283 [1.924 to 3.077]
  1 hour post bypass | 1.670 [1.334 to 2.383] | 2.068 [1.399 to 2.665]
  2 hour post bypass | 2.173 [1.898 to 2.507] | 2.201 [1.591 to 2.915]
  4 hour post bypass | 2.395 [2.237 to 2.988] | 3.116 [2.157 to 4.450]
  6 hour post bypass | 2.627 [2.320 to 3.317] | 3.485 [2.421 to 4.633]
  8 hour post bypass | 2.744 [2.454 to 3.369] | 3.143 [2.520 to 4.079]
  24 hour post bypass | 1.900 [1.550 to 2.901] | 2.269 [1.688 to 3.541]

4. Primary Outcome: The Examine and Measure Urinary NGAL to Measure Kidney Injury
Description: Urinary NGAL,a biomarker for kidney injury was measured.
Time Frame: A change in urinary NGAL 2 hours after bypass was stopped and 5 minutes after the start of spontaneous circulation was resumed.
Population: randomized as outlined in protocol
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Nesiritide | Placebo
Number analyzed (Participants) | 14 | 15
ng/ml | 124.566 [29.819 to 340.163] | 33.766 [9.825 to 425.434]

ADVERSE EVENTS:
Time Frame: June 2010 to December 2012
Arm/Group | Nesiritide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 3/15
Other Adverse Events (participants affected / at risk) | 2/14 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nesiritide (N=14) | Placebo (N=15)
Syncope (General disorders) | 0 (0) | 1 (1) — Subject went to the emergency room with a complaint of Syncope. Had surgery for an aortic valve replacement.
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Subject was hospitalized for Atrial Fibrillation.
Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient expired from respiratory insufficiency and failure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nesiritide (N=14) | Placebo (N=15)
Mediastinal exploration with evacuation of mediastinal and right clots/blood (Surgical and medical procedures) | 1 (1) | 0 (0) — Mediastinal exploration with evacuation of mediastinal and right clots/blood
Chest pain/ dysphagia (Cardiac disorders) | 1 (1) | 0 (0) — substernal chest pain and dysphagia
Shotness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — post operative visit, admitted due to increased shortness of breath.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No